CLINICAL TRIAL: NCT00087750
Title: Interaction Between IV Cocaine and Quetiapine
Brief Title: Interaction Between Cocaine and Quetiapine - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-MDS-0001-1
Record Dates: First submitted 2004-07-13; First posted 2004-07-16 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-03

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The purpose of this study is to assess the safety of intravenous (IV) cocaine in subjects taking quetiapine at 3 dosage levels.

DETAILED DESCRIPTION:
A placebo-controlled, double-blind, inpatient assessment of interaction between intravenous cocaine and quetiapine (seroquel) in cocaine-experienced subjects. To assess the safety of IV cocaine in subjects taking quetiapine at 3 dosage levels.

ELIGIBILITY:
Inclusion Criteria:

Includes but is not limited to: non-treatment seeking individuals. Must meet DSM-IV criteria for cocaine abuse or dependence. Must be able to verbalize understanding of consent and provide written informed consent and verbalize willingness to complete study procedures. Site will provide further details.

Exclusion Criteria:

Please contact site for further information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-10

PRIMARY OUTCOMES:
Adverse events
pharmacokinetic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Domenic Ciraulo, M.D., Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States